CLINICAL TRIAL: NCT01424917
Title: Noninvasive Predictors of Transplant Vasculopathy
Acronym: CAV
Status: Withdrawn | Type: Observational
Why Stopped: Investigator Left university
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0802M27524
Record Dates: First submitted 2011-03-22; First posted 2011-08-29 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Cardiac Allograft Vasculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Transplant: Heart Transplant subjects

SUMMARY:
Post transplant vasculopathy is a major negative outcome in heart transplantation. Current methods of detection are highly invasive and pose a risk to transplant recipients. Noninvasive markers of endothelial function can be used to detect transplant vasculopathy. Endothelial biomarkers such as: endothelial nitric oxide synthase, vascular cellular adhesion molecules, intracellular adhesion molecules, endothelin-1, thromboplastin, circulating endothelial cells, uric acid, and C-reactive play a role in the pathophysiologic mechanism of vasculopathy. Therefore, the investigators would like to assess the association between various endothelial biomarkers and the presence or absence of transplant vasculopathy.

DETAILED DESCRIPTION:
Cardiac transplantation has become the established treatment of choice for eligible patients with end-stage heart failure.

Cardiac allograft vasculopathy (CAV) is a major and potentially preventable limitation to long-term survival in cardiac transplant recipients. CAV affects up to 50% of recipients by year 5, though intimal thickening is present in up to 58% one year after transplantation. CAV is characterized by diffuse, concentric intimal hyperplasia, involving both epicardial and intramyocardial coronary arteries. In its most advanced stages, CAV is not amenable to standard revascularization procedures making the only cure re-transplantation. Given the limited donor pool and poor outcome, re-transplantation is not an option for all patients. CAV tends to be a silent process. Due to denervation of the transplanted heart, transplant recipients do not typically have chest pain, and thus the first symptoms of CAV may be those of heart failure or sudden cardiac death. Traditional risk factors are important in predicting the development of CAV, however non-traditional risk factors appear equally important and include cellular and humoral rejection, graft ischemia at the time of implantation, and cytomegalovirus (CMV). Despite the specific inciting event, the end result is endothelial dysfunction, which is the predecessor to CAV. Methods to detect, prevent, and treat endothelial dysfunction and subsequently CAV are few. The rapidity with which it develops, however, affords a great opportunity to study mechanisms and potential interventions in a relatively short period of time.

Chronic inflammation and immune activation and subsequent endothelial injury are felt to immunopathogenic in the development of CAV. Endothelial activation is a precursor to the development of transplant vasculopathy, and multiple biomarkers have been shown to correlate with the presence of endothelial dysfunction in transplant vasculopathy. (fig. 1) Endothelial activation, as determined by the presence of adhesion molecules, begins hours after brain death in a donor. VCAM-1, e-selectin, and p-selectin are expressed early after brain death in the donor and are elevated throughout transplantation in the recipient as a response to injury in the donor heart. P-selectin and VCAM remain elevated while e-selectin gradually decrease over three months. There is data suggesting that p-selectin and VCAM remain elevated up to 2 years after transplantation, suggesting persistent inflammation and immune activation after transplant. Furthermore, nitric oxide is the principal mediator of protective effects on the endothelium. The nitric oxide pathway is essential in maintaining vascular integrity in cardiac recipients, and inhibition of this pathway accelerates intimal thickening and worsens endothelial function caused by rejection. Intimal thickening is a marker of endothelial dysfunction and a precursor to the development of CAV.

Thus, these markers and others involved in atherogenesis, remodeling, immune activation and endothelial activation, may provide a useful modality in predicting the presence of vasculopathy. In addition, studying various components of the process, eg. inflammation and injury, will provide much needed information regarding targets for therapy.

Noninvasive assessments of peripheral artery function have demonstrated correlation with coronary artery function and are useful modalities to assess risk for coronary artery disease. Pulse wave amplitude and hyperemic response, using digital tonometry, are measures of peripheral endothelial function and have been shown to correlate with coronary microvascular function. Abnormalities in the coronary microcirculation and macrocirculation precede the development of vasculopathy in heart transplant recipients. Other measures of peripheral endothelial function include arterial elasticity (measured using CV Profiler, HDI, inc.) and flow-mediated dilatation of the brachial artery (FMD). These studies are sensitive noninvasive predictors of coronary artery disease, though have not been tested widely in the transplanted population. The investigators will use these studies to characterize peripheral artery function in heart transplant recipients and to determine whether they will be useful adjuncts in evaluating patients at risk for transplant vasculopathy. The ability to predict the development of vasculopathy before it is present provides an opportunity to intervene by escalating or modifying therapy and an opportunity to possibly prevent CAV, a major limitation to longevity of transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Age 18 years and greater
* Cardiac transplant recipients who have been transplanted for more than one year

Exclusion Criteria:

* Chronic kidney disease stage 4 defined as GFR <30
* Acute Rejection grade 3A or greater
* Active Infection
* Re-transplant
* Multiorgan Transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Transplant Subjects
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Noninvasive measurement of endothelial function and presence of vasculopathy | 1 year
  assess the association between various endothelial biomarkers and the presence or absence of transplant vasculopathy in patients after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Monica Colvin-Adams, MD,MS, Principal Investigator — Cardiology, University of Minnesota
Locations (1):
- Cardiology Division, University of Minnesota, Minneapolis, Minnesota, United States